CLINICAL TRIAL: NCT04090996
Title: Ffects of A Dual-Task Intervention in Postural Control in Multiple Sclerosis Patients With Low Level of Disability
Brief Title: Effects of A Dual-Task Intervention in Postural Control in Multiple Sclerosis Patients
Acronym: MOCOGSEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I16037 (MOCOGSEP)
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DT patients (Experimental)
  Interventions: Diagnostic Test: Dual TAsk

INTERVENTIONS:
Diagnostic Test: Dual TAsk — Motor assessment includes:
  * posturographic examination in Single-task (ST) and Double-task (DT)
  * an analysis of ST and DT walking;
  * Timed Up and Go (TUG) performances in real (rTUG) and imagined (iTUG) versions;

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory autoimmune disease affecting the central nervous system. It is the leading cause of severe non-traumatic disability in young adults (20-40 years). It affects more than 540,000 individuals in Europe and around 2.8 million people worldwide. The etiology of MS remains unknown to date, but probably results from a genetic predisposition associated with environmental factors (vitamin D deficiency, tobacco, vaccines, stress, diet, ...). MS is a neurological disease in which demyelination and axonal loss lead to many symptoms such as fatigue, spasticity, decreased sensitivity, muscle weakness, balance disorders, oculomotor visuals.

The Expanded Disability Status Scale (EDSS), which is used to rate functional disorders in MS patients, tends to underestimate these neurological disorders, which are often present in the early stages of the disease and are an important issue. major in the management and evolution of the disease.

Recently, it has been shown that motor and cognitive disorders appear in the early stages of the disease, yet these functions are not systematically evaluated in the early stages of the disease. These isolated or associated disorders often lead to real difficulties in realizing everyday activities. Since this disease affects young people who still have a professional activity, it is important not to underestimate the presence of these functional and cognitive disorders.

It is therefore necessary to seek more precise means of evaluation to detect certain neurological disorders.

Thus, the evaluation of these functions participates in the follow-up of the patient and makes it possible to better apprehend the evolution of these disorders in MS.

The investigators will use the concept of double-task to measure and evaluate these functional and cognitive disorders.

The dual task (DT) , is defined by the simultaneous completion of two tasks, one called "primary" and the other called "secondary", for which the performance changes are measured. The dual task paradigms are based on the assumption that two concurrently performed tasks interfere if they use identical functional and / or brain subsystems. In the case of a paradigm involving walking and another task, the interference is based on the assumption of the joint play of attention. The primary task is then the "attentional" task and the secondary task is represented by walking. Observed inferences are changes in the performance of one or both tasks that are measured by comparing single and dual task performance.

The assessment of DT's capabilities would improve the early detection of motor disorders in MS patients. Early identification of postural instability would make it easier to target care and improve patient follow-up. Conducting work on the concept of DT would improve our knowledge of this paradigm in MS.

Finally, a better understanding of double-stained mechanisms in MS could offer training programs

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18 to 65 years old;
* relapsing-remitting MS (RR);
* able to hold the station standing 180s without a device assistance;
* Expanded Disability Status Scale <4;
* able to give informed consent to participate in this study ;
* without any push in the 60 days before the participation in this study (to be clinically stable);
* no change in the treatment of MS since at least 2 month.

Exclusion Criteria:

* acute illness other than MS during the past 60 days;
* neurological and psychiatric diseases, except the SEP ;
* orthopedic and rheumatological disorders that may affect the market ;
* visual acuity <7/10 for the best eye after correction visual;
* patient undergoing psychiatric care;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Oscillation rate | DAy 1
  The presence of postural instability is determined by a value of oscillation rate greater than 2 standard deviations from the mean of the healthy population used in this study

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Magy, MD, Principal Investigator — CHU Limoges
Locations (1):
- Neurologie, Limoges, France